CLINICAL TRIAL: NCT05313620
Title: Effect of Tofacitinib on Coagulation and Platelet Function, and Its Role in Thromboembolic Events
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIS-2021-JAKihemo
Record Dates: First submitted 2021-09-02; First posted 2022-04-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis; Thromboembolism
Keywords: ulcerative colitis; Tromboembolism; Coagulation; Platelet Function; Tofacitinib; JAK inhibitors; anti-TNF; Infliximab; Adalimumab; Golimumab
MeSH Terms: conditions — Colitis, Ulcerative; Thromboembolism; Thrombosis | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ulcerative colitis patients treated with tofacitinib (Experimental): Tofacitinib 5 mg/day oral per clinical practice
  Interventions: Drug: Tofacitinib
- Ulcerative colitis patients treated with an anti-TNFα drug (Active Comparator): Infliximab (Infusion 5mg/kg milligram(s)/Kilogram-Intravenous use) per clinical practice, or adalimumab (Subcutaneus 40 mg milligram(s)-subcutaneus) per clinical practice, or golimumab (subcutaneus 50 mg milligram(s)-subcutaneus) per clinical practice
  Interventions: Drug: Infliximab Adalimumab y Golimumab
- healthy controls (No Intervention)

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib 5 MG/day per clinical practice
  Arms: Ulcerative colitis patients treated with tofacitinib
Drug: Infliximab Adalimumab y Golimumab — Infliximab (Infusion 5mg/kg milligram(s)/Kilogram-Intravenous use) per clinical practice or adalimumab (Subcutaneus 40 mg milligram(s)-subcutaneus) per clinical practice or or golimumab (subcutaneus 50 mg milligram(s)-subcutaneus) per clinical practice.
  Arms: Ulcerative colitis patients treated with an anti-TNFα drug

SUMMARY:
Post-authorization, prospective and unicenter clinical trial, in which patients with UC will be included. The treatment with anti-TNFα (infliximab, adalimumab or golimumab) or JAK-inhibitors (tofacitinib) will be initiated by clinical practice and the choice will be made at the discretion of the investigator at the center where the patients will be recruited (Hospital Universitario de La Princesa). In the case of the group of patients treated with tofacitinib, the selection will be made following the action protocol implemented in our center, in which this drug is usually reserved for those cases refractory to anti-TNFα and/or vedolizumab. There will be no random assignment of treatment. The drugs will be used in the approved indications and conditions of use.

DETAILED DESCRIPTION:
BACKGROUND

Ulcerative colitis (UC) is a chronic pathology that causes inflammation of the colonic mucosa (1, 2). The most common symptoms include bloody diarrhea, abdominal pain, and urgent bowel movements, which has a great impact on the quality of life (3). The chronic course of this disease is characterized by alternating periods of relapse and remission (4). The prevalence of UC is relatively high, with a rate of 505 cases per 100,000 population in Europe and 249 cases per 100,000 population in North America (5). In terms of incidence, it is increasing rapidly due to industrialization and westernization of lifestyles (6). The EpiCOM study recorded an overall incidence of 8.2 cases/100,000 person-years of UC (7). In Spain, a recent multicenter study coordinated from our center, which includes 17 Autonomous Communities of the country, confirmed that the current incidence of UC is higher than previously described, with rates of 8 new cases per 100,000 person-years, approximately (8,9). The complexity, the social burden and the costs of treatment make this disease very relevant for health systems. Specifically, in Europe, the annual direct cost is estimated at 9,000 euros per patient (regardless of severity) and 10,000 euros for those cases with moderate to severe UC. The total economic burden of UC has been estimated at 8-15 billion dollars in the US and 12-29 billion euros in Europe (10). All of this underscores the strategic importance of UC to society, including patients and health systems.

The goal of drug treatment is to control inflammation to prevent the development of progressive intestinal damage and the onset of complications, so patients can achieve an optimal quality of life. Biological drugs are effective in maintaining clinical remission (11-13). However, approximately half of the patients treated do not reach remission with biological treatment (14-16). The reason for this reduced effectiveness is because therapies are administered based on empirical approaches due to the lack of prognostic biomarkers, adapting them according to the clinical evolution and complications of each case (17).

A novel treatment for these refractory cases is tofacitinib (Xeljanz®), a synthetic small molecule inhibitor of JAK kinases, which has been shown to be effective in treating UC (18). Tofacitinib has been recently approved by the European Medicines Agency (EMA) and the Food and Drug Administration (FDA). It is indicated for the treatment of rheumatoid arthritis and active psoriatic arthritis, as well as in the treatment of adult patients with moderate to severe UC who have had an insufficient response, a loss of response or have been intolerant to conventional treatment or biological therapy. The recommended dose for UC is 10 mg twice daily for induction for 8 weeks, followed by 5 mg twice daily for maintenance (19). A relevant aspect to consider of this drug is its oral administration, unlike biological therapies, which are prescribed intravenously or subcutaneously.

Despite these advantages, it has been observed that some patients treated with tofacitinib have a higher incidence of severe thromboembolic events, including dose dependent pulmonary embolism and deep vein thrombosis. Recent data from a randomized, post-authorization safety trial (A3921133) in patients with rheumatoid arthritis over 50 years of age and at least one cardiovascular risk factor, treated with tofacitinib 10 mg twice daily, have shown an increased risk of pulmonary embolism and overall mortality. The increased risk of pulmonary embolism was 5 times higher compared to patients treated with anti-TNFα. The incidence rates of pulmonary embolism for tofacitinib 10 mg twice daily, tofacitinib 5 mg twice daily, and anti- TNFα were 0.54 (95% CI, 0.32-0.87), 0.27 (0.12-0.52), and 0.09 (0.02-0.26) per 100 patient-years treated, respectively. Furthermore, mortality due to any cause in the tofacitinib 10 mg every 12-hour group was 2 times higher than the mortality of the groups treated with tofacitinib 5 mg twice daily and anti-TNFα. The incidence rates of deep vein thrombosis for tofacitinib 10 mg twice daily, tofacitinib 5 mg twice daily, and anti-TNFα were 0.38 (0.20-0.67), 0.30 (0.14-0.55), and 0.18 (0.07-0.39) per 100 patient-years, respectively (20). These results support the current recommendation for cautious use of tofacitinib in patients with high thromboembolic risk.

As a result of the serious consequences associated with pulmonary embolism and the uncertainty about the underlying mechanism, the "Advisory Committee for Risk Assessment in Pharmacovigilance" decided to evaluate the impact of these findings on the benefit-risk balance of tofacitinib in all authorized indications, as well as the dose of administration. Both FDA and EMA have recently issued new warnings recommending "against" prescribing tofacitinib 10 mg twice daily for maintenance treatment in patients with UC who have one or more of the following known risk factors for venous thromboembolism (advanced age, obesity, diabetes, hypertension smoking, medical history of deep vein thrombosis and pulmonary embolism, immobilization of myocardial infarction in the previous three months, heart failure, use of combined hormonal contraceptives or hormone replacement therapy, inherited clotting disorders, neoplasia), unless appropriate alternative treatment is not available (21,22). In addition, the recommendations established by AEMPS to health professionals include monitoring all patients undergoing treatment with tofacitinib for signs and symptoms suggestive of pulmonary embolism, instructing them to request medical assistance immediately if they experience such symptoms (23).

Regarding thromboembolic risk specifically in UC patients treated with tofacitinib, the results of a recent post-hoc analysis showed that during tofacitinib treatment one patient had venous thromboembolism [incidence rate, patients with events/100 patient-years: 0.04; (0.00-0.23)] and four had pulmonary embolism [0.16 (0.04- 0.41)] at a dose of 10 mg predominantly, with risk factors for venous thromboembolism (24). Although data concerning UC patients are still limited, the results of the above-mentioned clinical trial in rheumatoid arthritis are relevant for any therapeutic indication.

Other drugs that inhibit the JAK-STAT pathway, such as baricitinib, ruxolitinib, and upadacitinib, have also been associated with an increased incidence of venous thromboembolism. However, the mechanism leading to these events is not known (25). Therefore, a possible class effect of JAK inhibitors in the development of these events cannot be ruled out. Moreover, other JAK inhibitors (pefacitinib, filgotinib and pacritinib) are currently being studied in phase 3 clinical trials in rheumatoid arthritis, atopic dermatitis, Crohn's disease and myelofibrosis (26-28). Because safety data on these new drugs are very limited, both regulatory agencies and clinical researchers have shown great concern about their thromboembolic risk. Therefore, it is clear that new studies are required to evaluate the safety of these new drugs.

This is an utmost need is order to offer these drugs to patients under the safest circumstances.

In summary, the pathophysiological mechanism that leads to an increased thromboembolic event in patients treated with tofacitinib or other JAK inhibitors is not currently known. Therefore, despite being effective and rapid drugs, their use has been restricted, since it is not known what would be the effective preventive antiplatelet or anticoagulation treatment, for example, to avoid thromboembolic events in these patients. This not only affects tofacitinib but may also involve the other JAK inhibitor drugs that will be approved for inflammatory bowel disease (or for other diseases) in the future. In this line, our project has an ambitious objective: to characterize in-depth this adverse event by studying the alterations in haemostasis. To that aim, the effect of tofacitinib on the general haemostatic profile (i.e., coagulation, platelet aggregation and activation) will be studied in vivo in patients with UC in the short and long term (baseline, 3 and 12 month follow-up).

Finally, it is highly probable that from the results obtained in the present project significant advances will be achieved in the knowledge of the molecular mechanisms involved in the appearance of venous thromboembolism caused by exposure to tofacitinib. Therefore, this will allow, in clinical practice, to adopt effective pharmacological measures and facilitate prevention strategies to reduce the onset of these complications. Furthermore, it is expected that the results obtained can be extrapolated to other JAK inhibitor drugs of the same family, due to the possible class effect.

ELIGIBILITY:
Inclusion Criteria:

EX VIVO STUDY IN PATIENTS WITH UC

PATIENTS WITH UC:

* Over 18 years old.
* Diagnosis of UC according to the criteria of the European Crohn's and Colitis Organisation (ECCO).
* Previous treatments are allowed, provided they have remained stable for the past 3 months.
* In the case of patients with active UC, they should have endoscopic activity within 1 month of starting the treatment (Mayo endoscopic sub-index of ≥ 2).
* Women of childbearing age using contraceptive methods with an error rate <1% per year. Examples of contraceptive methods whose error rate is <1% per year are:

  1. Intrauterine device (IUD).
  2. Bilateral tubal occlusion.
  3. Couple with vasectomy.
  4. Sexual abstinence.

INDIVIDUALS WITHOUT UC:

* Over 18 years old.
* Subjects not diagnosed with UC, or other inflammatory allergic, malignant or autoimmune diseases.
* Women of childbearing age using contraceptive methods with an error rate <1% per year. Examples of contraceptive methods whose error rate is <1% per year are:

  1. Intrauterine device (IUD).
  2. Bilateral tubal occlusion.
  3. Couple with vasectomy.
  4. Sexual abstinence.

IN VIVO STUDY IN PATIENTS WITH UC

PATIENTS WITH UC:

* Over 18 years old.
* Diagnosis of UC according to the criteria of the European Crohn's and Colitis Organisation (ECCO).
* Have indication of treatment with anti-TNFα (infliximab, adalimumab or golimumab) o tofacitinib.
* Be the first received JAK-inhibitor or anti-TNFα with a given mechanism of action.
* Have endoscopic activity of UC within 1 month of starting the treatment (Mayo endoscopic sub-index of ≥ 2).
* Previous treatments (including corticosteroids and immunosuppressants) are allowed provided that they have been stable for the last 3 months before beginning treatment with JAK-inhibitor or anti-TNFα and that they are maintained at a stable dose for the duration of the study
* Women of childbearing age using contraceptive methods with an error rate <1% per year. Examples of contraceptive methods whose error rate is <1% per year are:

  1. Intrauterine device (IUD).
  2. Bilateral tubal occlusion.
  3. Couple with vasectomy.
  4. Sexual abstinence.

INDIVIDUALS WITHOUT UC:

* Over 18 years old.
* Subjects not diagnosed with UC, or other inflammatory, allergic, malignant or autoimmune diseases.
* Women of childbearing age using contraceptive methods with an error rate <1% per year. Examples of contraceptive methods whose error rate is <1% per year are:

  1. Intrauterine device (IUD).
  2. Bilateral tubal occlusion.
  3. Couple with vasectomy.
  4. Sexual abstinence.

Exclusion Criteria:

EX VIVO STUDY IN PATIENTS WITH UC

PATIENTS WITH UC:

* Under 18 years old.
* Immune-mediated disease, neoplasm or active infection.
* Pregnancy or lactation.
* Alcohol or drug abuse.
* Ostomy.
* Abdominal surgery in the last 6 months.
* Colectomy.
* Active infection with hepatitis B, C or HIV virus.
* Medical history of thromboembolic events.
* Treatment with anticoagulants, antiplatelets or other drugs that alter the coagulation.
* Use of combined hormonal contraceptives or hormone replacement therapy.
* Hereditary coagulation disorders.
* Refusal to give consent for participation in the study.

INDIVIDUALS WITHOUT UC:

* Under 18 years of age.
* Advanced chronic disease or any other pathology that prevents the monitoring of the protocol of this study.
* Pregnancy or lactation.
* Alcohol or drug abuse.
* Ostomy.
* Abdominal surgery in the last 6 months.
* Colectomy.
* Active infection with hepatitis B, C or HIV virus.
* Medical history of thromboembolic events.
* Treatment with anticoagulants, antiplatelets or other drugs that alter the coagulation.
* Use of combined hormonal contraceptives or hormone replacement therapy.
* Hereditary coagulation disorders.
* Refusal to give consent for participation in the study.

IN VIVO STUDY IN PATIENTS WITH UC

PATIENTS WITH UC:

* Under 18 years old.
* Immune-mediated disease.
* Neoplasm or active infection.
* Pregnancy or lactation.
* Alcohol or drug abuse.
* Ostomy.
* Colectomy.
* Active infection with hepatitis B, C or HIV virus.
* Indication of anti-TNFα or JAK-inhibitors treatment for a cause other than UC.
* Have previously received a drug with the same mechanism of action (anti-TNFα or JAK-inhibitors)
* Medical history of thromboembolic events.
* Treatment with anticoagulants, antiplatelets or other drugs that alter the coagulation.
* Use of combined hormonal contraceptives or hormone replacement therapy.
* Hereditary coagulation disorders.
* Refusal to give consent for participation in the study.

INDIVIDUALS WITHOUT UC:

* Under 18 years of age.
* Advanced chronic disease or any other pathology that prevents the monitoring of the protocol of this study.
* Pregnancy or lactation.
* Alcohol or drug abuse.
* Active infection with hepatitis B, C or HIV virus.
* Finding of macroscopic alterations during the colonoscopy or finding of relevant inflammatory alterations in the biopsies obtained during the colonoscopy.
* Treatment with immunomodulators, immunosuppressants, corticosteroids or other drugs that alter the immune system.
* Medical history of thromboembolic events.
* Treatment with anticoagulants, antiplatelets or other drugs that alter the coagulation.
* Use of combined hormonal contraceptives or hormone replacement therapy.
* Hereditary coagulation disorders.
* Refusal to give consent for participation in the study.
* Abdominal surgery in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
platelet activation | 1 year
  Platelet activation status will be assessed ex vivo in platelet-rich plasma (PRP) samples from UC patients (active and quiescent) and healthy controls incubated in the absence or presence of drug (tofacitinib or anti-TNFα). Regarding the in vivo study, platelet activation will be analyzed in samples from patients with active UC before and after initiating treatment with tofacitinib or anti-TNFα. It will be mesured by rate of platelet agregation

SECONDARY OUTCOMES:
Endoscopic activity | 1 year
  It will be evaluated by the Mayo endoscopic sub-score; endoscopic activity will be considered as ≥ 2.
Endoscopic response | 1 year
  It will be defined as a decrease of ≥ 1 point in the Mayo endoscopic sub-score 3 months after starting treatment.
Endoscopic remission | 1 year
  It will be defined as an endoscopic subscore ≤1, 3 months after starting treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ordas I, Eckmann L, Talamini M, Baumgart DC, Sandborn WJ. Ulcerative colitis. Lancet. 2012 Nov 3;380(9853):1606-19. doi: 10.1016/S0140-6736(12)60150-0. Epub 2012 Aug 20. PMID 22914296
- [Background] Hoivik ML, Moum B, Solberg IC, Henriksen M, Cvancarova M, Bernklev T; IBSEN Group. Work disability in inflammatory bowel disease patients 10 years after disease onset: results from the IBSEN Study. Gut. 2013 Mar;62(3):368-75. doi: 10.1136/gutjnl-2012-302311. Epub 2012 Jun 20. PMID 22717453
- [Background] Kornbluth A, Sachar DB; Practice Parameters Committee of the American College of Gastroenterology. Ulcerative colitis practice guidelines in adults: American College Of Gastroenterology, Practice Parameters Committee. Am J Gastroenterol. 2010 Mar;105(3):501-23; quiz 524. doi: 10.1038/ajg.2009.727. Epub 2010 Jan 12. PMID 20068560
- [Background] Ye Y, Pang Z, Chen W, Ju S, Zhou C. The epidemiology and risk factors of inflammatory bowel disease. Int J Clin Exp Med. 2015 Dec 15;8(12):22529-42. eCollection 2015. PMID 26885239
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Burisch J, Pedersen N, Cukovic-Cavka S, Brinar M, Kaimakliotis I, Duricova D, Shonova O, Vind I, Avnstrom S, Thorsgaard N, Andersen V, Krabbe S, Dahlerup JF, Salupere R, Nielsen KR, Olsen J, Manninen P, Collin P, Tsianos EV, Katsanos KH, Ladefoged K, Lakatos L, Bjornsson E, Ragnarsson G, Bailey Y, Odes S, Schwartz D, Martinato M, Lupinacci G, Milla M, De Padova A, D'Inca R, Beltrami M, Kupcinskas L, Kiudelis G, Turcan S, Tighineanu O, Mihu I, Magro F, Barros LF, Goldis A, Lazar D, Belousova E, Nikulina I, Hernandez V, Martinez-Ares D, Almer S, Zhulina Y, Halfvarson J, Arebi N, Sebastian S, Lakatos PL, Langholz E, Munkholm P; EpiCom-group. East-West gradient in the incidence of inflammatory bowel disease in Europe: the ECCO-EpiCom inception cohort. Gut. 2014 Apr;63(4):588-97. doi: 10.1136/gutjnl-2013-304636. Epub 2013 Apr 20. PMID 23604131
- [Background] Chaparro M, Barreiro-de Acosta M, Benitez JM, Cabriada JL, Casanova MJ, Ceballos D, Esteve M, Fernandez H, Ginard D, Gomollon F, Lorente R, Nos P, Riestra S, Rivero M, Robledo P, Rodriguez C, Sicilia B, Torrella E, Garre A, Garcia-Esquinas E, Rodriguez-Artalejo F, Gisbert JP; EpidemIBD study group of GETECCU. EpidemIBD: rationale and design of a large-scale epidemiological study of inflammatory bowel disease in Spain. Therap Adv Gastroenterol. 2019 May 21;12:1756284819847034. doi: 10.1177/1756284819847034. eCollection 2019. PMID 31205485
- [Background] Cohen RD, Yu AP, Wu EQ, Xie J, Mulani PM, Chao J. Systematic review: the costs of ulcerative colitis in Western countries. Aliment Pharmacol Ther. 2010 Apr;31(7):693-707. doi: 10.1111/j.1365-2036.2010.04234.x. Epub 2010 Jan 11. PMID 20064142
- [Background] Ungaro R, Mehandru S, Allen PB, Peyrin-Biroulet L, Colombel JF. Ulcerative colitis. Lancet. 2017 Apr 29;389(10080):1756-1770. doi: 10.1016/S0140-6736(16)32126-2. Epub 2016 Dec 1. PMID 27914657
- [Background] Chaparro M, Garre A, Ricart E, Iborra M, Mesonero F, Vera I, Riestra S, Garcia-Sanchez V, Luisa De Castro M, Martin-Cardona A, Aldeguer X, Minguez M, de-Acosta MB, Rivero M, Munoz F, Andreu M, Bargallo A, Gonzalez-Munoza C, Perez Calle JL, Garcia-Sepulcre MF, Bermejo F, Huguet JM, Cabriada JL, Gutierrez A, Manosa M, Villoria A, Carbajo AY, Lorente R, Garcia-Lopez S, Piqueras M, Hinojosa E, Arajol C, Sicilia B, Conesa AM, Sainz E, Almela P, Llao J, Roncero O, Camo P, Taxonera C, Domselaar MV, Pajares R, Legido J, Madrigal R, Lucendo AJ, Alcain G, Domenech E, Gisbert JP; GETECCU study group. Short and long-term effectiveness and safety of vedolizumab in inflammatory bowel disease: results from the ENEIDA registry. Aliment Pharmacol Ther. 2018 Oct;48(8):839-851. doi: 10.1111/apt.14930. PMID 30281832
- [Background] Sands BE, Sandborn WJ, Panaccione R, O'Brien CD, Zhang H, Johanns J, Adedokun OJ, Li K, Peyrin-Biroulet L, Van Assche G, Danese S, Targan S, Abreu MT, Hisamatsu T, Szapary P, Marano C; UNIFI Study Group. Ustekinumab as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2019 Sep 26;381(13):1201-1214. doi: 10.1056/NEJMoa1900750. PMID 31553833
- [Background] Ford AC, Sandborn WJ, Khan KJ, Hanauer SB, Talley NJ, Moayyedi P. Efficacy of biological therapies in inflammatory bowel disease: systematic review and meta-analysis. Am J Gastroenterol. 2011 Apr;106(4):644-59, quiz 660. doi: 10.1038/ajg.2011.73. Epub 2011 Mar 15. PMID 21407183
- [Background] Danese S, Allez M, van Bodegraven AA, Dotan I, Gisbert JP, Hart A, Lakatos PL, Magro F, Peyrin-Biroulet L, Schreiber S, Tarabar D, Vavricka S, Halfvarson J, Vermeire S. Unmet Medical Needs in Ulcerative Colitis: An Expert Group Consensus. Dig Dis. 2019;37(4):266-283. doi: 10.1159/000496739. Epub 2019 Feb 6. PMID 30726845
- [Background] Gordon JP, McEwan PC, Maguire A, Sugrue DM, Puelles J. Characterizing unmet medical need and the potential role of new biologic treatment options in patients with ulcerative colitis and Crohn's disease: a systematic review and clinician surveys. Eur J Gastroenterol Hepatol. 2015 Jul;27(7):804-12. doi: 10.1097/MEG.0000000000000378. PMID 25933126
- [Background] Gisbert JP, Chaparro M. Predictors of Primary Response to Biologic Treatment [Anti-TNF, Vedolizumab, and Ustekinumab] in Patients With Inflammatory Bowel Disease: From Basic Science to Clinical Practice. J Crohns Colitis. 2020 Jun 19;14(5):694-709. doi: 10.1093/ecco-jcc/jjz195. PMID 31777929
- [Background] Chaparro M, Garre A, Mesonero F, Rodriguez C, Barreiro-de Acosta M, Martinez-Cadilla J, Arroyo MT, Mancenido N, Sierra-Ausin M, Vera-Mendoza I, Casanova MJ, Nos P, Gonzalez-Munoza C, Martinez T, Bosca-Watts M, Calafat M, Busquets D, Girona E, Llao J, Martin-Arranz MD, Piqueras M, Ramos L, Suris G, Bermejo F, Carbajo AY, Casas-Deza D, Fernandez-Clotet A, Garcia MJ, Ginard D, Gutierrez-Casbas A, Hernandez L, Lucendo AJ, Marquez L, Merino-Ochoa O, Rancel FJ, Taxonera C, Lopez Sanroman A, Rubio S, Domenech E, Gisbert JP. Tofacitinib in Ulcerative Colitis: Real-world Evidence From the ENEIDA Registry. J Crohns Colitis. 2021 Jan 13;15(1):35-42. doi: 10.1093/ecco-jcc/jjaa145. PMID 32969471
- [Background] Coskun M, Salem M, Pedersen J, Nielsen OH. Involvement of JAK/STAT signaling in the pathogenesis of inflammatory bowel disease. Pharmacol Res. 2013 Oct;76:1-8. doi: 10.1016/j.phrs.2013.06.007. Epub 2013 Jul 2. PMID 23827161
- [Background] Sandborn WJ, Panes J, Sands BE, Reinisch W, Su C, Lawendy N, Koram N, Fan H, Jones TV, Modesto I, Quirk D, Danese S. Venous thromboembolic events in the tofacitinib ulcerative colitis clinical development programme. Aliment Pharmacol Ther. 2019 Nov;50(10):1068-1076. doi: 10.1111/apt.15514. Epub 2019 Oct 9. PMID 31599001
- [Background] Scott IC, Hider SL, Scott DL. Thromboembolism with Janus Kinase (JAK) Inhibitors for Rheumatoid Arthritis: How Real is the Risk? Drug Saf. 2018 Jul;41(7):645-653. doi: 10.1007/s40264-018-0651-5. PMID 29500799
- [Background] Sands BE, Sandborn WJ, Feagan BG, Lichtenstein GR, Zhang H, Strauss R, Szapary P, Johanns J, Panes J, Vermeire S, O'Brien CD, Yang Z, Bertelsen K, Marano C; Peficitinib-UC Study Group. Peficitinib, an Oral Janus Kinase Inhibitor, in Moderate-to-severe Ulcerative Colitis: Results From a Randomised, Phase 2 Study. J Crohns Colitis. 2018 Nov 9;12(10):1158-1169. doi: 10.1093/ecco-jcc/jjy085. PMID 29917064
- [Background] van der Heijde D, Baraliakos X, Gensler LS, Maksymowych WP, Tseluyko V, Nadashkevich O, Abi-Saab W, Tasset C, Meuleners L, Besuyen R, Hendrikx T, Mozaffarian N, Liu K, Greer JM, Deodhar A, Landewe R. Efficacy and safety of filgotinib, a selective Janus kinase 1 inhibitor, in patients with active ankylosing spondylitis (TORTUGA): results from a randomised, placebo-controlled, phase 2 trial. Lancet. 2018 Dec 1;392(10162):2378-2387. doi: 10.1016/S0140-6736(18)32463-2. Epub 2018 Oct 22. PMID 30360970
- [Background] Mesa RA, Vannucchi AM, Mead A, Egyed M, Szoke A, Suvorov A, Jakucs J, Perkins A, Prasad R, Mayer J, Demeter J, Ganly P, Singer JW, Zhou H, Dean JP, Te Boekhorst PA, Nangalia J, Kiladjian JJ, Harrison CN. Pacritinib versus best available therapy for the treatment of myelofibrosis irrespective of baseline cytopenias (PERSIST-1): an international, randomised, phase 3 trial. Lancet Haematol. 2017 May;4(5):e225-e236. doi: 10.1016/S2352-3026(17)30027-3. Epub 2017 Mar 20. PMID 28336242
- [Background] Piran S, Schulman S. Management of venous thromboembolism: an update. Thromb J. 2016 Oct 4;14(Suppl 1):23. doi: 10.1186/s12959-016-0107-z. eCollection 2016. PMID 27766049
- [Background] Kyrle PA, Rosendaal FR, Eichinger S. Risk assessment for recurrent venous thrombosis. Lancet. 2010 Dec 11;376(9757):2032-9. doi: 10.1016/S0140-6736(10)60962-2. Epub 2010 Dec 3. PMID 21131039
- [Background] Danese S, Sans M, Fiocchi C. Inflammatory bowel disease: the role of environmental factors. Autoimmun Rev. 2004 Jul;3(5):394-400. doi: 10.1016/j.autrev.2004.03.002. PMID 15288007
- [Background] Giannotta M, Tapete G, Emmi G, Silvestri E, Milla M. Thrombosis in inflammatory bowel diseases: what's the link? Thromb J. 2015 Apr 2;13:14. doi: 10.1186/s12959-015-0044-2. eCollection 2015. PMID 25866483
- [Background] Montoro-Garcia S, Schindewolf M, Stanford S, Larsen OH, Thiele T. The Role of Platelets in Venous Thromboembolism. Semin Thromb Hemost. 2016 Apr;42(3):242-51. doi: 10.1055/s-0035-1570079. Epub 2016 Feb 29. PMID 26926584
- [Background] Monroe DM, Hoffman M, Roberts HR. Platelets and thrombin generation. Arterioscler Thromb Vasc Biol. 2002 Sep 1;22(9):1381-9. doi: 10.1161/01.atv.0000031340.68494.34. PMID 12231555
- [Background] Bergmeier W, Hynes RO. Extracellular matrix proteins in hemostasis and thrombosis. Cold Spring Harb Perspect Biol. 2012 Feb 1;4(2):a005132. doi: 10.1101/cshperspect.a005132. PMID 21937733
- [Background] Fernandez-Bello I, Lopez-Longo FJ, Arias-Salgado EG, Jimenez-Yuste V, Butta NV. Behcet's disease: new insight into the relationship between procoagulant state, endothelial activation/damage and disease activity. Orphanet J Rare Dis. 2013 May 27;8:81. doi: 10.1186/1750-1172-8-81. PMID 23711081
- [Background] Alvarez-Roman MT, Fernandez-Bello I, Jimenez-Yuste V, Martin-Salces M, Arias-Salgado EG, Rivas Pollmar MI, Justo Sanz R, Butta NV. Procoagulant profile in patients with immune thrombocytopenia. Br J Haematol. 2016 Dec;175(5):925-934. doi: 10.1111/bjh.14412. Epub 2016 Oct 21. PMID 27766635
- [Background] Ozdemir ZC, Duzenli Kar Y, Gunduz E, Turhan AB, Bor O. Evaluation of hypercoagulability with rotational thromboelastometry in children with iron deficiency anemia. Hematology. 2018 Oct;23(9):664-668. doi: 10.1080/10245332.2018.1452456. Epub 2018 Mar 15. PMID 29544395
- [Background] Coelho MC, Vieira Neto L, Kasuki L, Wildemberg LE, Santos CV, Castro G, Gouvea G, Veloso OC, Gadelha T, Gadelha MR. Rotation thromboelastometry and the hypercoagulable state in Cushing's syndrome. Clin Endocrinol (Oxf). 2014 Nov;81(5):657-64. doi: 10.1111/cen.12491. Epub 2014 Jun 12. PMID 24815846
- [Background] Mulder MB, Proctor KG, Valle EJ, Livingstone AS, Nguyen DM, Van Haren RM. Hypercoagulability After Resection of Thoracic Malignancy: A Prospective Evaluation. World J Surg. 2019 Dec;43(12):3232-3238. doi: 10.1007/s00268-019-05123-7. PMID 31407092
- [Background] Campello E, Spiezia L, Zabeo E, Maggiolo S, Vettor R, Simioni P. Hypercoagulability detected by whole blood thromboelastometry (ROTEM(R)) and impedance aggregometry (MULTIPLATE(R)) in obese patients. Thromb Res. 2015 Mar;135(3):548-53. doi: 10.1016/j.thromres.2015.01.003. Epub 2015 Jan 7. PMID 25592651
- [Background] Bedreli S, Straub K, Achterfeld A, Willuweit K, Katsounas A, Saner F, Wedemeyer H, Herzer K. The Effect of Immunosuppression on Coagulation After Liver Transplantation. Liver Transpl. 2019 Jul;25(7):1054-1065. doi: 10.1002/lt.25476. Epub 2019 May 30. PMID 31021493
- [Background] Grant AL, Letson HL, Morris JL, McEwen P, Hazratwala K, Wilkinson M, Dobson GP. Tranexamic acid is associated with selective increase in inflammatory markers following total knee arthroplasty (TKA): a pilot study. J Orthop Surg Res. 2018 Jun 18;13(1):149. doi: 10.1186/s13018-018-0855-5. PMID 29914535
- [Background] Brophy DF, Martin EJ, Christian Barrett J, Nolte ME, Kuhn JG, Gerk PM, Carr ME, Pelzer H, Agerso H, Ezban M, Hedner U. Monitoring rFVIIa 90 mug kg(-)(1) dosing in haemophiliacs: comparing laboratory response using various whole blood assays over 6 h. Haemophilia. 2011 Sep;17(5):e949-57. doi: 10.1111/j.1365-2516.2011.02492.x. Epub 2011 Mar 1. PMID 21362113
- [Background] Tsantes AE, Kyriakou E, Ikonomidis I, Katogiannis K, Papadakis I, Douramani P, Kopterides P, Kapsimali V, Lekakis J, Tsangaris I, Bonovas S. Comparative Assessment of the Anticoagulant Activity of Rivaroxaban and Dabigatran in Patients With Nonvalvular Atrial Fibrillation: A Noninterventional Study. Medicine (Baltimore). 2016 Apr;95(14):e3037. doi: 10.1097/MD.0000000000003037. PMID 27057830
- [Background] Patel-Hett S, Martin EJ, Mohammed BM, Rakhe S, Sun P, Barrett JC, Nolte ME, Kuhn J, Pittman DD, Murphy JE, Brophy DF. Marstacimab, a tissue factor pathway inhibitor neutralizing antibody, improves coagulation parameters of ex vivo dosed haemophilic blood and plasmas. Haemophilia. 2019 Sep;25(5):797-806. doi: 10.1111/hae.13820. Epub 2019 Jul 23. PMID 31336410
- [Background] Yada K, Nogami K, Ogiwara K, Shida Y, Furukawa S, Yaoi H, Takeyama M, Kasai R, Shima M. Global coagulation function assessed by rotational thromboelastometry predicts coagulation-steady state in individual hemophilia A patients receiving emicizumab prophylaxis. Int J Hematol. 2019 Oct;110(4):419-430. doi: 10.1007/s12185-019-02698-8. Epub 2019 Jun 28. PMID 31254165
- [Background] Walden K, Shams Hakimi C, Jeppsson A, Karlsson M. Effects of fibrinogen supplementation on clot formation in blood samples from cardiac surgery patients before and after tranexamic acid administration. Transfus Med. 2019 Oct;29(5):319-324. doi: 10.1111/tme.12604. Epub 2019 May 22. PMID 31115109
- [Background] Lillemae K, Laine AT, Schramko A, Niemi TT. Effect of Albumin in Combination With Mannitol on Whole-blood Coagulation In Vitro Assessed by Thromboelastometry. J Neurosurg Anesthesiol. 2018 Jul;30(3):265-272. doi: 10.1097/ANA.0000000000000438. PMID 28498140
- [Background] Lak M, Scharling B, Blemings A, Sharifian R, Maleki Z, Daraee A, Arjmand AR, Hedner U. Evaluation of rFVIIa (NovoSeven) in Glanzmann patients with thromboelastogram. Haemophilia. 2008 Jan;14(1):103-10. doi: 10.1111/j.1365-2516.2007.01592.x. Epub 2007 Dec 7. PMID 18070065
- [Background] Wang Y, Andrews M, Yang Y, Lang S, Jin JW, Cameron-Vendrig A, Zhu G, Reheman A, Ni H. Platelets in thrombosis and hemostasis: old topic with new mechanisms. Cardiovasc Hematol Disord Drug Targets. 2012 Dec;12(2):126-32. doi: 10.2174/1871529x11202020126. PMID 23030445
- [Background] Berndt MC, Metharom P, Andrews RK. Primary haemostasis: newer insights. Haemophilia. 2014 May;20 Suppl 4:15-22. doi: 10.1111/hae.12427. PMID 24762270
- [Background] Mackman N. Triggers, targets and treatments for thrombosis. Nature. 2008 Feb 21;451(7181):914-8. doi: 10.1038/nature06797. PMID 18288180
- [Background] Gurbel PA, Bliden K, Barnett SD, Witt C, Zou H, Tantry U. An Ex Vivo Study to Evaluate the Effect of Tegaserod on Platelet Activation and Aggregation. J Cardiovasc Pharmacol Ther. 2021 Jan;26(1):40-50. doi: 10.1177/1074248420942004. Epub 2020 Jul 16. PMID 32672062
- [Background] Meah MN, Raftis J, Wilson SJ, Perera V, Garonzik SM, Murthy B, Everlof JG, Aronson R, Luettgen J, Newby DE. Antithrombotic Effects of Combined PAR (Protease-Activated Receptor)-4 Antagonism and Factor Xa Inhibition. Arterioscler Thromb Vasc Biol. 2020 Nov;40(11):2678-2685. doi: 10.1161/ATVBAHA.120.314960. Epub 2020 Sep 10. PMID 32907366
- [Background] Cirillo P, Taglialatela V, Pellegrino G, Morello A, Conte S, Di Serafino L, Cimmino G. Effects of colchicine on platelet aggregation in patients on dual antiplatelet therapy with aspirin and clopidogrel. J Thromb Thrombolysis. 2020 Aug;50(2):468-472. doi: 10.1007/s11239-020-02121-8. PMID 32335777
- [Background] Alvarez Roman MT, Fernandez Bello I, Arias-Salgado EG, Rivas Pollmar MI, Jimenez Yuste V, Martin Salces M, Butta NV. Effects of thrombopoietin receptor agonists on procoagulant state in patients with immune thrombocytopenia. Thromb Haemost. 2014 Jul 3;112(1):65-72. doi: 10.1160/TH13-10-0873. Epub 2014 Feb 6. PMID 24500066
- [Background] Lee J, Jung CW, Jeon Y, Kim TK, Cho YJ, Koo CH, Choi YH, Kim KB, Hwang HY, Kim HR, Park JY. Effects of preoperative aspirin on perioperative platelet activation and dysfunction in patients undergoing off-pump coronary artery bypass graft surgery: A prospective randomized study. PLoS One. 2017 Jul 17;12(7):e0180466. doi: 10.1371/journal.pone.0180466. eCollection 2017. PMID 28715503
- [Background] Vrigkou E, Tsangaris I, Bonovas S, Kopterides P, Kyriakou E, Konstantonis D, Pappas A, Anthi A, Gialeraki A, Orfanos SE, Armaganidis A, Tsantes A. Platelet and coagulation disorders in newly diagnosed patients with pulmonary arterial hypertension. Platelets. 2019;30(5):646-651. doi: 10.1080/09537104.2018.1499890. Epub 2018 Jul 26. PMID 30047809
- [Background] Peyrin-Biroulet L, Sandborn W, Sands BE, Reinisch W, Bemelman W, Bryant RV, D'Haens G, Dotan I, Dubinsky M, Feagan B, Fiorino G, Gearry R, Krishnareddy S, Lakatos PL, Loftus EV Jr, Marteau P, Munkholm P, Murdoch TB, Ordas I, Panaccione R, Riddell RH, Ruel J, Rubin DT, Samaan M, Siegel CA, Silverberg MS, Stoker J, Schreiber S, Travis S, Van Assche G, Danese S, Panes J, Bouguen G, O'Donnell S, Pariente B, Winer S, Hanauer S, Colombel JF. Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE): Determining Therapeutic Goals for Treat-to-Target. Am J Gastroenterol. 2015 Sep;110(9):1324-38. doi: 10.1038/ajg.2015.233. Epub 2015 Aug 25. PMID 26303131
- [Background] Kamm MA, Sandborn WJ, Gassull M, Schreiber S, Jackowski L, Butler T, Lyne A, Stephenson D, Palmen M, Joseph RE. Once-daily, high-concentration MMX mesalamine in active ulcerative colitis. Gastroenterology. 2007 Jan;132(1):66-75; quiz 432-3. doi: 10.1053/j.gastro.2006.10.011. Epub 2006 Oct 12. PMID 17241860
- [Background] Van Assche G, Sandborn WJ, Feagan BG, Salzberg BA, Silvers D, Monroe PS, Pandak WM, Anderson FH, Valentine JF, Wild GE, Geenen DJ, Sprague R, Targan SR, Rutgeerts P, Vexler V, Young D, Shames RS. Daclizumab, a humanised monoclonal antibody to the interleukin 2 receptor (CD25), for the treatment of moderately to severely active ulcerative colitis: a randomised, double blind, placebo controlled, dose ranging trial. Gut. 2006 Nov;55(11):1568-74. doi: 10.1136/gut.2005.089854. Epub 2006 Apr 7. PMID 16603634
- [Background] D'Haens G, Feagan B, Colombel JF, Sandborn WJ, Reinisch W, Rutgeerts P, Carbonnel F, Mary JY, Danese S, Fedorak RN, Hanauer S, Lemann M; International Organization for Inflammatory Bowel Diseases (IOIBD) and the Clinical Trial Committee Clincom of the European Crohn's and Colitis Organisation (ECCO). Challenges to the design, execution, and analysis of randomized controlled trials for inflammatory bowel disease. Gastroenterology. 2012 Dec;143(6):1461-9. doi: 10.1053/j.gastro.2012.09.031. Epub 2012 Sep 20. PMID 23000597
- [Background] Nunes T, Barreiro-de Acosta M, Nos P, Marin-Jimenez I, Bermejo F, Ceballos D, Iglesias E, Gomez-Senent S, Torres Y, Ponferrada A, Arevalo JA, Hernandez V, Calvet X, Ginard D, Monfort D, Chaparro M, Mancenido N, Dominguez-Antonaya M, Villalon C, Perez-Calle JL, Munoz C, Nunez H, Carpio D, Aramendiz R, Bujanda L, Estrada-Oncins S, Hermida C, Barrio J, Casis MB, Duenas-Sadornil MC, Fernandez L, Calvo-Cenizo MM, Botella B, de Francisco R, Ayala E, Sans M; RECLICU Study Group of GETECCU. Usefulness of oral beclometasone dipropionate in the treatment of active ulcerative colitis in clinical practice: the RECLICU Study. J Crohns Colitis. 2010 Dec;4(6):629-36. doi: 10.1016/j.crohns.2010.07.003. PMID 21122572